CLINICAL TRIAL: NCT00948233
Title: Combating Tobacco Use in the United States Army
Brief Title: Project COMBAT: Combating Tobacco Use in the United States Army
Status: Withdrawn | Type: Observational
Why Stopped: Military related changes led to to no initiation of recruitment.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2009-0222; W81XWH-09-2-0033 (Other: DOD)
Record Dates: First submitted 2009-07-16; First posted 2009-07-29 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Smoking; Smoking Cessation
Keywords: Tobacco; Smoking Cessation; Prevention; Smokeless tobacco; Habit
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use; Habits | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples at the 12-month follow-up visit to measure level of cotinine, a chemical related to tobacco use.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention: Educational video game
  Interventions: Behavioral: Video Game; Behavioral: Surveys
- Standard Care: Pamphlets on stopping tobacco use
  Interventions: Behavioral: Pamphlet; Behavioral: Surveys

INTERVENTIONS:
Behavioral: Video Game — Educational anti-tobacco video game played on arcade-type kiosk for three 30-minute sessions, plus CD-ROM disc of game to use as needed, and series of illustrated materials to go along with computer sessions.
  Groups: Intervention
Behavioral: Pamphlet — Self-help pamphlet about stopping and avoiding tobacco use, provided by the National Institutes of Health.
  Groups: Standard Care
Behavioral: Surveys — Computer surveys taken at 4 points throughout the study.
  Other Names: Questionnaire

SUMMARY:
The goal of this behavioral research study is to test a new multimedia anti-tobacco video game tailored to the U.S. Army. Researchers want to study how using the program affects tobacco use in soldiers, as compared to standard anti-tobacco programs.

DETAILED DESCRIPTION:
Researchers in the M. D. Anderson Department of Behavioral Science are developing a new video game program for young U.S. Army service members. The game addresses stopping and preventing the use of cigarettes and smokeless tobacco. Soldiers (ages 18-35 years) stationed at Fort Hood, Texas, who are not scheduled to be mobilized for a 13-month period, will be invited to take part in the study.

The Study Groups:

If you choose to take part in this study, you will be assigned to a type of study intervention. The personnel companies on-base have been randomly assigned (as in the flip of a coin) to offer participating service members 1 of the following 2 programs: either the educational video game (called the "intervention"), or pamphlets on stopping tobacco use (called "standard care"). Each company will receive only 1 of the 2 programs, and all participating service members in the same company will receive the same program. Each company has an equal chance of being assigned to either program.

Intervention:

Participants in the intervention group will have a month to use the educational anti-tobacco video game located in areas that will provide convenient access. The game will be made available using an arcade-type kiosk which houses the computer game. After playing the video game on the kiosk for three 30-minute sessions, you will then be given a CD-ROM disc of the game to use as needed. After finishing these three 30-minute computer sessions, you will also receive a series of printed materials that go along with the computer sessions.

Standard Care:

The standard care participants will receive a self-help pamphlet about stopping and avoiding tobacco use, provided by the National Institutes of Health.

Both Intervention and Standard Care Groups:

No matter which group your company is assigned to, if you choose to take part, you will be asked to complete surveys by computer at 4 points throughout the study. The survey will include questions about tobacco use, such as how much tobacco you use, how many times you have tried to quit, how ready you are to quit, how dependent you are on nicotine, any withdrawal and breathing symptoms you experience, your level of alcohol use, and support from family and friends. Each survey should take about 30 minutes to complete.

The first surveys will take place at the start of study participation. The intervention group will complete the second survey right after finishing the program. The standard care group will complete this second survey at about the same time as the intervention group. Both groups will also complete the third and fourth surveys at 6- and 12-month follow-ups.

You will be asked to provide saliva samples at the 12-month follow-up visit. Researchers will use these saliva samples to measure the level of cotinine, a chemical in your saliva that is related to tobacco use. You will be asked to spit into a clean plastic container. A dipstick will be placed in the container for at least 30 minutes. After reading the dipstick and recording the result, the study staff will throw away the saliva sample right away.

You will also be told about the nicotine replacement therapy and other tobacco cessation services available at no cost through the Carl R. Darnall Army Medical Center (CRDAMC) Tobacco Cessation Program at Fort Hood. M. D. Anderson is collaborating with the CRDAMC Tobacco Cessation Program on this study.

This is an investigational study. Up to 2050 soldiers will be asked to take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty service members, age 18 or above, who have entered the Army stationed at Joint Base San Antonio
2. Does not have to be a current smoker or user of alternative tobacco products
3. Must provide contact information including: an address, telephone number, and an email address
4. Willing to answer two questions regarding status of smoking and smokeless tobacco use on study survey
5. Have access to the Internet
6. Speak, read and write in English at a sixth-grade literacy level

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Soldiers stationed at Fort Hood, Texas, who are not scheduled to be mobilized for a 13-month period.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Reductions in Smoking Initiation/Smokeless Tobacco Use and Smoking Cessation | Baseline, immediately following completion of the program, and at 6- and 12-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Alex Prokhorov, MD, PHD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org